CLINICAL TRIAL: NCT07353866
Title: Effectiveness of Combination of Square Stepping Exercise and Bosu Ball Exercise on Postural Sway, and Biomotor Abilities in Badminton Players
Brief Title: Role of Stepping and BOSU Ball Training in Enhancing Postural Balance and Performance of Badminton Players
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: INTI International University (Other)
Collaborators: Saveetha University (Other)
Responsible Party: Principal Investigator, Vinosh Kumar Purushothaman, Lecturer, INTI International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: INTI IUFHLSRCBPHTI1NY12024/018
Record Dates: First submitted 2026-01-11; First posted 2026-01-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Sports Injury; Injury Prevention in Sports
Keywords: Postural stability; Balance; Health risk; Lower limb explosive power; Square Stepping exercise
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Square stepping and BOSU ball exercise group (Experimental): Square stepping and BOSU ball exercise group will receive Square Stepping Exercise and BOSU ball training for the period of 8 weeks, 3 times per week.
  Interventions: Other: Square stepping + BOSU ball exercise
- BOSU ball and Shadow training group (Experimental): BOSU ball and Shadow training group receives BOSU ball training Protocol along with shadow training for the period of 8 weeks, 3 days per week
  Interventions: Other: BOSU ball and Shadow training
- Conventional Exercise group (Placebo Comparator): Conventional Exercise group will undergo regular conventional badminton training for the period of 8 weeks, 3 days per week
  Interventions: Other: Conventional Training

INTERVENTIONS:
Other: Square stepping + BOSU ball exercise — Participants in Square Stepping Exercise and BOSU ball exercise group will perform both Square Stepping Exercise and BOSU ball training. Square Stepping Exercise will be implemented on Monday, Wednesday and Friday for a period of 8 weeks, each session lasts for 30 minutes. Meanwhile, all participants in this group will undergo specified BOSU ball protocol on Tuesday Thursday and Saturday for the same duration of 8 weeks, 30 minutes each session. The Square Stepping training comprises of a series of forward, backward, lateral, and diagonal steps, with the complexity of pattern increasing from week 2 to week 8.
  Arms: Square stepping and BOSU ball exercise group
Other: BOSU ball and Shadow training — Participants in BOSU ball and Shadow training group will perform both BOSU ball and Shadow training. BOSU ball will be implemented on 3 days a week for a period of 8 weeks, each session lasts for 30 minutes. Meanwhile, all participants in this group will undergo Shadow training on 3 days a week for a period of 8 weeks, each session lasts for 30 minutes.
  Arms: BOSU ball and Shadow training group
Other: Conventional Training — Participants in the conventional training group will undergo regular training for the period of 8 weeks, 3 session in a week each session last for 50-60 minutes.
  Arms: Conventional Exercise group

SUMMARY:
Influence of Square Stepping and BOSU Ball Exercise on Lower Extremity Balance and Strength in Badminton Players: An Expanded Explanation for Patients, Families, and Health Care Providers

Badminton is a dynamic and physically demanding sport that requires a unique combination of speed, agility, balance, coordination, and muscular strength. Unlike many other sports, badminton involves frequent and rapid changes in direction, explosive lunges, sudden stops, jumps, and controlled landings, often performed repeatedly within a short period of time. These movements place significant stress on the lower extremities, particularly the ankles, knees, hips, and surrounding muscles. As a result, maintaining good balance and adequate lower limb strength is essential not only for optimal performance but also for injury prevention.

This research study focuses on understanding how two specific exercise methods, Square Stepping Exercise (SE) and BOSU Ball Exercise (BE)-can influence lower extremity balance and strength when used together in badminton players. While each of these exercises has already been shown to provide benefits when used individually, their combined effect, particularly in relation to badminton-specific physical demands, has not been well explored. The findings of this study may help athletes, families, coaches, physiotherapists, and other health care providers make informed decisions about training, rehabilitation, and injury prevention strategies.

Understanding the Physical Demands of Badminton To appreciate the importance of this study, it is essential to understand the physical demands of badminton. Badminton is often underestimated as a recreational sport; however, at both competitive and recreational levels, it is one of the fastest racket sports in the world. Players must react quickly to the shuttlecock, which can travel at extremely high speeds, and move efficiently across the court using complex footwork patterns.

Key physical requirements of badminton include:

Dynamic balance, which allows players to maintain body control while moving, lunging, jumping, or landing. Lower limb strength, especially in the quadriceps, hamstrings, calf muscles, and hip muscles, to generate power and absorb forces. Agility and coordination, enabling quick directional changes and precise foot placement. Postural control to stabilize the body during rapid and asymmetrical movements. During a typical rally, a badminton player may perform multiple lunges, side steps, backward steps, and jumps within seconds. These movements are often performed on one leg, increasing the challenge to balance and joint stability. If a player lacks adequate balance or strength, they may struggle to control these movements efficiently, which can negatively affect performance and increase the likelihood of injury.

Common Lower Extremity Injuries in Badminton:

Because of the sport's high physical demands, badminton players are at risk of various lower extremity injuries. These injuries can occur due to overuse, improper landing mechanics, muscle weakness, or poor balance control. Common injuries include:

Ankle sprains are often caused by sudden changes in direction or unstable landings. Knee injuries, such as patellar tendinopathy or ligament strain Muscle strains, particularly in the quadriceps, hamstrings, and calf muscles Overuse injuries, resulting from repetitive movements without adequate recovery. Many of these injuries are linked to deficits in balance, muscle strength, and neuromuscular control. Improving these physical components through targeted exercise programs is therefore a key focus of sports training and rehabilitation.

In badminton, exercises that improve balance and lower limb strength can help players move more efficiently, react faster, and maintain stability during challenging movements. Balance and strength training also improve communication between the nervous system and muscles, which is essential for precise and controlled movements.

Square Stepping Exercise (SE) is a structured form of stepping activity performed on a grid or pattern marked on the floor, usually consisting of multiple squares arranged in rows and columns. Participants are instructed to step into specific squares in a particular sequence, moving forward, backward, sideways, or diagonally. A BOSU ball is a training device consisting of a half-sphere dome attached to a flat base.

While square stepping and BOSU ball exercises are effective individually, they target balance and strength in slightly different ways. Square stepping focuses more on movement accuracy, coordination, and directional control, whereas BOSU ball exercise emphasizes stability, muscle activation, and joint control under unstable conditions. Combining these two exercises may improve both static and dynamic balance and enhance functional strength relevant to badminton movement efficiency.

DETAILED DESCRIPTION:
Badminton is a highly dynamic and physically demanding racket sport that requires players to demonstrate an exceptional blend of speed, agility, balance, coordination, and muscular strength throughout play. Unlike many sports that involve predictable movement patterns or longer pauses between actions, badminton is characterized by rapid rallies, sudden changes in direction, explosive lunges, quick accelerations and decelerations, repeated jumps, and controlled single-leg landings, all performed within very short time frames. These movements place considerable mechanical and neuromuscular demands on the body, particularly on the lower extremities, including the ankles, knees, hips, and the surrounding muscles and connective tissues. Each lunge, jump, or pivot requires the lower limb joints to absorb and generate force efficiently while maintaining stability and alignment. Consequently, maintaining adequate balance and lower limb strength is not only fundamental for optimal performance in badminton but is also essential for reducing the risk of injury and ensuring long-term participation in the sport. When balance or strength is compromised, even slightly, players may experience reduced movement efficiency, delayed reactions, poor landing mechanics, and increased joint stress, all of which can negatively impact performance and safety.

The present research study focuses on understanding how two specific exercise approaches-Square Stepping Exercise and BOSU Ball Exercise -influence lower extremity balance and strength when applied together in badminton players. Both of these exercise methods have independently demonstrated positive effects on balance, strength, coordination, and neuromuscular control in various populations, including athletes and individuals undergoing rehabilitation. However, despite their individual effectiveness, the combined or synergistic impact of these exercises, particularly in relation to the unique physical and movement demands of badminton, has not been sufficiently explored. By examining the influence of a combined square stepping and BOSU ball exercise program, this study aims to fill an important gap in sports science and rehabilitation research. The findings of this research may provide valuable insights for badminton players seeking to enhance performance, families who support athletes in maintaining health and safety, coaches who design training programs, and health care providers such as physiotherapists and sports trainers who are involved in injury prevention and rehabilitation.

To fully appreciate the importance of this study, it is necessary to understand the specific physical demands of badminton and how they challenge the body. Badminton is often perceived as a recreational or leisure activity; however, at both competitive and recreational levels, it is recognized as one of the fastest racket sports in the world. The shuttlecock can travel at extremely high speeds, requiring players to react almost instantaneously and move efficiently across the court using complex footwork patterns. These footwork patterns involve repeated forward lunges, lateral movements, backward stepping, rapid turns, and vertical jumps, often performed in unpredictable sequences. Players are required to maintain precise control of their body position while responding to visual cues and executing technically demanding strokes, all of which place a high demand on balance, coordination, and muscular strength.

Dynamic balance is a critical physical requirement in badminton, as it allows players to maintain body control while moving, lunging, jumping, and landing, often on a single leg. Unlike static balance, which involves maintaining stability in a fixed position, dynamic balance requires continuous adjustments of the body's center of mass over a changing base of support. In badminton, these adjustments must occur rapidly and repeatedly during play. Lower limb strength is equally important, particularly in the quadriceps, hamstrings, calf muscles, and hip muscles, as these muscle groups generate the force needed for powerful movements and absorb the impact forces associated with jumping and landing. Adequate strength in these muscles helps protect the joints from excessive stress and supports efficient movement patterns. Agility and coordination enable players to change direction quickly and place their feet accurately during fast rallies, while postural control allows the trunk and pelvis to remain stable during rapid and asymmetrical movements. Together, these physical attributes contribute to effective performance and injury resilience in badminton.

During a typical rally, a badminton player may perform several lunges, side steps, backward movements, and jumps within a matter of seconds. Many of these movements are executed on one leg, which significantly increases the demand on balance and joint stability. Single-leg activities require precise neuromuscular control to maintain alignment of the ankle, knee, and hip while managing external forces. If a player lacks adequate balance, strength, or neuromuscular coordination, controlling these movements becomes more challenging. This can result in inefficient movement patterns, slower reaction times, reduced accuracy in stroke execution, and increased stress on the joints and soft tissues. Over time, these deficits may contribute to fatigue, performance decline, and a higher risk of injury.

Due to the high physical demands of badminton, players are susceptible to a range of lower extremity injuries. These injuries may occur as a result of overuse, improper landing mechanics, muscle weakness, poor balance control, or inadequate recovery between training sessions and matches. Ankle sprains are among the most common injuries in badminton and often occur during sudden changes in direction or unstable landings after jumps. Knee injuries, including patellar tendinopathy, ligament strains, and cartilage stress, are also frequently reported due to repetitive loading, deep lunges, and rapid deceleration movements. Muscle strains, particularly in the quadriceps, hamstrings, and calf muscles, may occur when muscles are unable to cope with the high forces generated during explosive movements. Additionally, overuse injuries can develop when repetitive movements are performed without sufficient rest, leading to cumulative tissue stress. Many of these injuries are closely linked to deficits in balance, muscle strength, and neuromuscular control, highlighting the importance of targeted exercise programs in sports training and rehabilitation.

Exercise interventions that specifically address balance and lower limb strength play a crucial role in improving movement efficiency, enhancing performance, and reducing injury risk in badminton players. Balance training helps players develop better control of their body position during complex movements, while strength training enhances the muscles' ability to generate and absorb force. Importantly, balance and strength training also improve communication between the nervous system and the muscles, a process known as neuromuscular adaptation. This improved communication allows muscles to respond more quickly and appropriately to changes in movement and loading conditions, which is essential for precise and controlled actions during badminton play.

Square Stepping Exercise is one such training method that has gained attention for its ability to improve balance, coordination, and lower limb control. Square stepping is a structured form of stepping activity performed on a grid or pattern marked on the floor, typically consisting of multiple squares arranged in rows and columns. Participants are instructed to step into specific squares in predetermined sequences, moving forward, backward, sideways, or diagonally. These stepping patterns require individuals to focus on foot placement accuracy, timing, and directional changes, all of which are highly relevant to badminton footwork. Square stepping exercises can be progressively modified by increasing the complexity or speed of the stepping patterns, making them suitable for athletes of different skill levels. Through repeated practice, square stepping helps improve dynamic balance, coordination, reaction time, and lower limb control, which are essential for efficient movement on the badminton court.

BOSU ball exercise represents another effective training approach, particularly for enhancing balance and strength under unstable conditions. A BOSU ball is a training device consisting of a half-sphere dome attached to a flat base, creating an unstable surface that challenges the body's balance system. Exercises performed on a BOSU ball require continuous adjustments by the muscles and joints to maintain stability, thereby increasing muscle activation and joint control. BOSU ball exercises can be performed in various positions, including standing, squatting, lunging, and jumping, and can involve one or both legs. These exercises are commonly used in sports training and physiotherapy to improve postural control, joint stability, muscle strength, and neuromuscular coordination. For badminton players, BOSU ball exercises can simulate the unstable conditions experienced during sudden stops, landings, and directional changes, helping the body adapt to the demands of the sport.

While square stepping and BOSU ball exercises are effective when used independently, they target balance and strength through slightly different mechanisms. Square stepping primarily emphasizes movement accuracy, coordination, directional control, and cognitive engagement, as participants must remember and execute specific stepping sequences. In contrast, BOSU ball exercise places greater emphasis on stability, muscle activation, and joint control under unstable conditions. By combining these two exercise methods, it is possible to address both the movement-based and stability-based components of balance and strength. This combined approach may lead to improvements in both static and dynamic balance, enhance functional strength relevant to badminton movements, and improve overall movement efficiency.

The rationale for combining square stepping and BOSU ball exercises lies in their complementary effects on the neuromuscular system. Square stepping trains the ability to move efficiently through space with accurate foot placement, while BOSU ball exercises train the ability to maintain stability when the base of support is unstable. Together, these exercises may provide a more comprehensive stimulus for improving balance, strength, and coordination in badminton players. Improved balance and strength may allow players to perform movements with greater confidence, control, and efficiency, thereby enhancing performance and reducing the risk of injury.

In summary, badminton is a sport that places high physical demands on the lower extremities, requiring a combination of balance, strength, agility, and coordination. Deficits in these areas can negatively affect performance and increase injury risk. Square stepping and BOSU ball exercises are two training methods that have demonstrated benefits in improving balance and strength through different mechanisms. By exploring the combined influence of these exercises on lower extremity balance and strength in badminton players, this study aims to provide valuable evidence to support effective training, rehabilitation, and injury prevention strategies. The findings may benefit athletes striving for better performance, families seeking to support healthy participation in sports, and health care providers designing evidence-based exercise programs tailored to the specific demands of badminton.

ELIGIBILITY:
Inclusion Criteria:

* minimum of 1 year of experience in badminton
* competed in a minimum of 2 club-level badminton tournaments in the past 6 months

Exclusion Criteria:

* any lower limb surgery
* ACL injury, or any other injury in the lower extremity in the past 1 year
* involved any other form of physical training other than badminton-specific training
* neurological disorders that may affect the balance and proprioception

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-01-21 (Estimated); Primary Completion 2026-06-24 (Estimated); Study Completion 2026-08-21 (Estimated)

PRIMARY OUTCOMES:
Postural Sway | From enrollment to the end of treatment at 8 weeks
  Postural sway refers to the small, continuous movements of the body that occur while a person is standing upright and attempting to maintain balance. One widely used and cost-effective tool for this purpose is the Wii Balance Board. Originally developed for gaming, the Wii Balance Board has been validated for use as a force platform in scientific and clinical research. It contains four pressure sensors positioned at each corner of the board, which measure vertical ground reaction forces generated by the user. When a person stands on the board, changes in weight distribution across the sensors are recorded, allowing the calculation of the center of pressure (COP).

SECONDARY OUTCOMES:
Vertical Jump Height | From enrollment to the end of treatment at 8 weeks
  To assess standing reach height, the participant will be asked to stand next to a wall and reach upward as high as possible, marking the highest point reached on the wall with chalk. The participant will then stand 10 cm away from the wall to allow free arm movement. With the fingers coated in chalk, the participant will be instructed to perform a countermovement by bending the knees and swinging the arms backward, then jump and reach upward as high as possible to mark the wall. The vertical jump height will be determined by calculating the difference between the standing reach mark and the highest jump mark on the wall.

CONTACTS AND LOCATIONS:
Overall Officials: Vinosh Kumar Purushothaman, Principal Investigator — INTI International University; Vinodhkumar Ramalingam, Study Director — Saveetha College of Physiotherapy
Locations (1):
- University Badminton Club, Seremban, Negeri Sembilan, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) will not be shared because the data collected contain personal and potentially identifiable information related to participants' health, physical performance, and assessment results. Sharing IPD could compromise participant privacy and confidentiality, which were assured during the informed consent process.

REFERENCES:
- [Background] Clark RA, Mentiplay BF, Pua YH, Bower KJ. Reliability and validity of the Wii Balance Board for assessment of standing balance: A systematic review. Gait Posture. 2018 Mar;61:40-54. doi: 10.1016/j.gaitpost.2017.12.022. Epub 2017 Dec 30. PMID 29304510
- [Background] Lu Z, Zhou L, Gong W, Chuang S, Wang S, Guo Z, Bao D, Zhang L, Zhou J. The Effect of 6-Week Combined Balance and Plyometric Training on Dynamic Balance and Quickness Performance of Elite Badminton Players. Int J Environ Res Public Health. 2022 Jan 30;19(3):1605. doi: 10.3390/ijerph19031605. PMID 35162627
- [Background] Wang YH, Liu YH, Yang YR, Wang RY. Effects of square-stepping exercise on motor and cognitive function in older adults - A systematic review and meta-analysis. Geriatr Nurs. 2021 Nov-Dec;42(6):1583-1593. doi: 10.1016/j.gerinurse.2021.10.022. Epub 2021 Nov 10. PMID 34773911
- [Background] Malwanage KT, Senadheera VV, Dassanayake TL. Effect of balance training on footwork performance in badminton: An interventional study. PLoS One. 2022 Nov 17;17(11):e0277775. doi: 10.1371/journal.pone.0277775. eCollection 2022. PMID 36395192